CLINICAL TRIAL: NCT05022173
Title: Helmet NIV Versus Facemask NIV in Acute Respiratory Failure: A Pilot Randomized Control Trial
Brief Title: Helmet NIV in Acute Respiratory Failure
Acronym: HELMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13412
Record Dates: First submitted 2021-07-26; First posted 2021-08-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Failure
Keywords: non-invasive ventilation; Helmet non-invasive ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helmet NIV (Experimental): Patients randomized to the intervention arm will receive NIV through a phthalate free helmet (CaStar, STARMED) via an ICU ventilator in pressure support (PS) mode.
  Interventions: Device: Helmet Non-Invasive Ventilation
- Facemask NIV (Active Comparator): Patients in the control arm will be randomized to the traditional facemask interface. The facemask group will use the same ICU ventilator being used for the helmet group.
  Interventions: Device: Facemask Non-Invasive Ventilation

INTERVENTIONS:
Device: Helmet Non-Invasive Ventilation — The helmet interface is a modality which is used to deliver NIV to patients with respiratory failure. A transparent hood is placed over the entire head of the patient with a seal at the neck using a soft collar.
  Arms: Helmet NIV
Device: Facemask Non-Invasive Ventilation — The facemask interface is a modality which is also used to deliver NIV to patients with respiratory failure. A large mask covering the mouth and nose is strapped to the patient's face to create a seal.
  Arms: Facemask NIV

SUMMARY:
Non-invasive ventilation (NIV) is a form of respiratory support that has been shown to prevent invasive mechanical ventilation and reduce mortality. This study will investigate the feasibility of performing a larger study examining whether a new modality of NIV, the helmet, is superior to the current face mask in reducing mortality in patients with sudden respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients who are admitted to the adult ICU
* 2) deemed to require NIV, as per the clinical team, for acute respiratory failure.

Exclusion Criteria:

* 1) with impending cardiac arrest or need for intubation
* 2) Glasgow coma scale <9
* 3) tracheostomy or upper airway obstruction
* 4) elevated intracranial pressure
* 5) untreated pneumothorax
* 6) who refuse endotracheal intubation (do not intubate order documented)
* 7) facial trauma
* 8) are unable to wear the helmet or facemask
* 9) who use NIV chronically

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Consent Rate | 1 year
  Percentage of patients or SDMs approached for consent who give consent
Recruitment Rate | 1 year
  Number of patients recruited to the study per centre
Protocol adherence percentage | 1 year
  Adherence to pre-specified fixed protocol on how helmet interface is implemented (settings, weaning etc.) Any protocol deviations will be recorded and marked as protocol non-adherence.

SECONDARY OUTCOMES:
Endotracheal intubation | 28 days
  Number of patients requiring endotracheal intubation
ICU mortality | 28 days
  Number of patients who die in ICU
Hospital mortality | 60 days
  Number of patients who die in hospital
ICU length of stay | Censored at 28 days
  Number of days that each patient spends in ICU
Hospital length of stay | Censored at 60 days
  Number of days that each patients spends in hospital
Duration of non-invasive ventilation | Censored at 28 days
  Number of days that patient receives non-invasive ventilation
Duration of invasive ventilation | Censored at 28 days
  Number of days that patient receives invasive ventilation
Adverse events | 28 days
  Any complications related to NIV use
Comfort | 28 days
  Patient comfort with non-invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Bram Rochwerg, MD, Principal Investigator — Hamilton Health Science
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided